CLINICAL TRIAL: NCT03435640
Title: A Phase 1/2, Open-label, Multicenter, Dose Escalation and Dose Expansion Study of NKTR-262 in Combination With Bempegaldesleukin (NKTR-214) With or Without Nivolumab in Patients With Locally Advanced or Metastatic Solid Tumor Malignancies
Brief Title: REVEAL Study of NKTR-262 in Combination With NKTR-214 and Nivolumab in Patients With Locally Advanced / Metastatic Solid Tumor Malignancies
Acronym: REVEAL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Based on the overall results from the Phase 1 part of the study the sponsor decided to end the study. The decision was not due to safety reasons.
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-262-01; 2018-004625-84 (EudraCT Number)
Record Dates: First submitted 2018-02-06; First posted 2018-02-19 (Actual); Results first posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Melanoma; Merkel Cell Carcinoma; Triple Negative Breast Cancer; Head and Neck Squamous Cell Carcinoma; Renal Cell Carcinoma; Colorectal Cancer; Sarcoma
Keywords: Bempegaldesleukin (NKTR-214); NKTR-262; Nivolumab; Opdivo®; Metastatic; Locally advanced; Relapsed/Refractory; TLR7/8; CD122
MeSH Terms: conditions — Melanoma; Carcinoma, Merkel Cell; Triple Negative Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Colorectal Neoplasms; Sarcoma; Neoplasm Metastasis; Recurrence | interventions — bempegaldesleukin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NKTR-262 + bempegaldesleukin or + bempegaldesleukin with nivolumab (Experimental): Phase 1: NKTR-262 in escalating doses, combined with bempegaldesleukin. The goal of this dose escalation part of the study is to establish a recommended Phase 1b dose for NKTR-262 + bempegaldesleukin with nivolumab, followed by a dose-confirmation cohort.
  Interventions: Drug: NKTR-262; Drug: bempegaldesleukin; Drug: nivolumab

INTERVENTIONS:
Drug: NKTR-262 — During Phase 1 Doublet: Patients receive escalating doses of NKTR-262 IT (starting dose 0.03 mg) in 3-week treatment cycles. During Phase 1 Doublet (Cohort A), Phase 2 Doublet: Patients were to receive the RP2D of NKTR-262.
  During Phase 1 Triplet (Cohort B), and Phase 2 Triplet: Patients receive the RP2D of NKTR-262.
Drug: bempegaldesleukin — During Phase 1 Doublet (Cohort A), and proposed Phase 2 Doublet: Patients receive 0.006 mg/kg bempegaldesleukin administered in 3-week treatment cycles.
  During Phase 1 Triplet (Cohort B), and proposed Phase 2 Triplet: Patients receive 0.006 mg/kg bempegaldesleukin administered in 3-week treatment cycles.
  Other Names: NKTR-214
Drug: nivolumab — During Phase 1 Triplet (Cohort B), and proposed Phase 2 Triplet: Patients receive a nivolumab flat dose of 360 mg administered in 3-week treatment cycles.
  Other Names: Opdivo®

SUMMARY:
Patients received intratumoral (IT) injections of NKTR-262 in 3-week cycles for up to 3 cycles; bempegaldesleukin with or without nivolumab was administered every 3 weeks (q3w), and treatment continued until unacceptable toxicity, death, or disease progression per RECIST 1.1. Based on Phase 1 results of the study, the decision was made not to start the Phase 2 part of the study and the study was terminated.

DETAILED DESCRIPTION:
Cancer treatments that couple pharmacological activation of tumor antigen presentation with activation and expansion of CD8+ T and natural killer (NK) cells in the tumor environment have the potential to induce an effective anti-tumor immune response in patients. NKTR-262 is a small molecule agonist of toll-like receptors (TLRs) 7/8 designed to be retained in the tumor micro-environment in order to activate antigen-presenting cells (APC), such as dendritic cells, to create new antigen-specific cytotoxic T cells. As a CD122-biased agonist, bempegaldesleukin monotherapy increases newly proliferative CD8+ T cells in tumors. NKTR-262 plus bempegaldesleukin is expected to increase expansion of antigen-specific CD8+ T cells. In preclinical studies, a single IT injection of NKTR-262 plus IV bempegaldesleukin resulted in complete abscopal effects in tumor models. Preliminary clinical data show bempegaldesleukin plus nivolumab enhances immune-stimulatory responses. The REVEAL trial will assess safety and anti-tumor activity of NKTR-262 with bempegaldesleukin +/- nivolumab for the treatment of selected cancers.

* Melanoma (1st-line and relapsed/refractory)
* Merkel Cell Carcinoma (2nd-line and relapsed/refractory)
* Triple Negative Breast Cancer (1st- and 2nd-line and relapsed/refractory)
* Renal Cell Carcinoma (1st-line and relapsed/refractory)
* Colorectal Cancer (2nd-line and relapsed/refractory; MSI non-high)
* Colorectal Cancer (2nd 3rd-line+, I-O therapy naive; relapsed/refractory; MSI high)
* Head and Neck Squamous Cell Carcinoma (2nd-line and relapsed/refractory)
* Sarcoma (2nd-line and relapsed/refractory)

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of a locally advanced (not amenable to curative therapy such as surgical resection) metastatic cancer of the following histologies: melanoma (MEL), Merkel cell carcinoma (MCC), triple-negative breast cancer (TNBC), renal cell carcinoma (RCC), colorectal cancer, head and neck squamous cell carcinoma (HNSCC), or sarcoma.
* Life expectancy > 12 weeks as determined by the Investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Measurable disease per RECIST 1.1.
* Patients enrolled in Cohorts 1-10, Cohort A, Cohort B and Phase 2 Doublet must be refractory to all therapies known to confer clinical benefit to their disease.
* Fresh tumor tissue available for cellular characterization and programmed cell death protein 1 (PD-L1) status.
* Injected lesions (up to two) must be between 20 mm and 90 mm in diameter for IT injection; lesions must be accessible for baseline and on-treatment biopsies. Any liver lesion targeted for injection must not exceed 50 mm at the time of injection.
* Demonstrated adequate organ function within 14 days of Cycle 1 Day 1 (C1D1).

Key Exclusion Criteria:

* Use of an investigational agent or an investigational device within 21 days before administration of first dose of study drug(s).
* Patients treated with prior interleukin-2 (IL-2).
* Patients who have been previously treated with a toll-like receptor (TLR) agonist (excluding topical agents) and patients who have received experimental cancer vaccines.
* Patients who have received systemic interferon (IFN)α within the previous 6 months prior to enrollment to the study.
* Other active malignancy, except non-melanomic skin cancer
* Evidence of clinically significant interstitial lung disease or active, noninfectious pneumonitis.
* Prior surgery or radiotherapy within 14 days of initiating study drug(s). Patients must have recovered from all radiation-related toxicities, not required corticosteroids and have not had radiation pneumonitis.
* Prolonged Fridericia's corrected QT interval (QTcF) > 450 ms for men and > 470 ms for women at Screening.

History of unstable or deteriorating cardiac disease within the previous 6 months prior to screening including but not limited to the following:

* Unstable angina or myocardial infarction.
* Congestive heart failure (NYHA Class III or IV).
* Uncontrolled clinically significant arrhythmias.
* Patients with a history of any retinal disorders (e.g., retinal detachment, diabetic retinopathy, retinal hemorrhage, macular degeneration).
* Uveal melanoma will be excluded
* Patients with tumor that invade the superior vena cava or other major blood vessels.

Additional general and tumor specific inclusion and exclusion criteria will apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (14):
- United States (14):
  - HonorHealth, Scottsdale, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Center, Emory University Hospital, Atlanta, Georgia
  - University of Kansas Research Center, Fairway, Kansas
  - Henry Ford Health System, Detroit, Michigan
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rolig AS, Rose DC, McGee GH, Rubas W, Kivimae S, Redmond WL. Combining bempegaldesleukin (CD122-preferential IL-2 pathway agonist) and NKTR-262 (TLR7/8 agonist) improves systemic antitumor CD8+ T cell cytotoxicity over BEMPEG+RT. J Immunother Cancer. 2022 Apr;10(4):e004218. doi: 10.1136/jitc-2021-004218. PMID 35444059

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 NKTR-262 (0.03 mg) + Bempegaldesleukin (Administered Staggered): Phase 1 (dose escalation) Cohort 1 Patients received NKTR-262 intratumorally at 0.03 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) (administered staggered [Day 3] in Cycles 2-3).
  The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort 2 NKTR-262 (0.06 mg) + Bempegaldesleukin (Administered Staggered): Phase 1 (dose escalation) Cohort 2 Patients received NKTR-262 intratumorally at 0.06 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) (administered staggered [Day 3] in Cycles 2-3).
  The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort 3 NKTR-262 (0.06 mg) + Bempegaldesleukin (Administered the Same Day): Phase 1 (dose escalation) Cohort 3 Patients received NKTR-262 intratumorally at 0.06 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) administered on the same day.
  The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort 4 NKTR-262 (0.12 mg) + Bempegaldesleukin (Administered the Same Day): Phase 1 (dose escalation) Cohort 4 Patients received NKTR-262 intratumorally at 0.12 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) administered on the same day.
  The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort 5 NKTR-262 (0.24 mg) + Bempegaldesleukin (Administered the Same Day): Phase 1 (dose escalation) Cohort 5 Patients received NKTR-262 intratumorally at 0.24 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) administered on the same day.
  The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort 6 NKTR-262 (0.48 mg) + Bempegaldesleukin (Administered the Same Day): Phase 1 (dose escalation) Cohort 6 Patients received NKTR-262 intratumorally at 0.48 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) administered on the same day.
  The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort 7 NKTR-262 (0.96 mg) + Bempegaldesleukin (Administered the Same Day): Phase 1 (dose escalation) Cohort 7 Patients received NKTR-262 intratumorally at 0.96 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) administered on the same day.
  The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort 8 NKTR-262 (1.92 mg) + Bempegaldesleukin (Administered the Same Day): Phase 1 (dose escalation) Cohort 8 Patients received NKTR-262 intratumorally at 1.92 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) administered on the same day.
  The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort 9 NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day): Phase 1 (dose escalation) Cohort 9 Patients received NKTR-262 intratumorally at 3.84 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) administered on the same day.
  The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort A NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day): Cohort A explored same-day administration of NKTR-262 intratumorally at the RP2D (3.84 mg) and bempegaldesleukin IV (0.006 mg/kg) q3w.
- Cohort B NKTR-262 (3.84 mg) + Bempegaldesleukin + Nivolumab: Cohort B explored same-day administration of NKTR-262 intratumorally at the RP2D (3.84 mg) and bempegaldesleukin IV (0.006 mg/kg) q3w plus nivolumab IV (360 mg) q3w, starting in Cycle 1.
Period: Overall Study
Arm/Group | Cohort 1 NKTR-262 (0.03 mg) + Bempegaldesleukin (Administered Staggered) | Cohort 2 NKTR-262 (0.06 mg) + Bempegaldesleukin (Administered Staggered) | Cohort 3 NKTR-262 (0.06 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 4 NKTR-262 (0.12 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 5 NKTR-262 (0.24 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 6 NKTR-262 (0.48 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 7 NKTR-262 (0.96 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 8 NKTR-262 (1.92 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 9 NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort A NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort B NKTR-262 (3.84 mg) + Bempegaldesleukin + Nivolumab
Started | 3 | 3 | 4 | 3 | 4 | 4 | 4 | 3 | 8 | 14 | 14
Completed | 3 | 2 | 3 | 1 | 4 | 4 | 1 | 3 | 8 | 12 | 11
Not Completed | 0 | 1 | 1 | 2 | 0 | 0 | 3 | 0 | 0 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 9 NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day): Phase 1 (dose escalation) Cohort 9 Patients received NKTR-262 intratumorally at 3.84 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) administered on the same day.The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort A NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day): Cohort A explored same-day administration of NKTR-262 at the RP2D (3.84 mg) and bempegaldesleukin (0.006 mg/kg) q3w.
- Cohort B NKTR-262 (3.84 mg) + Bempegaldesleukin + Nivolumab: Cohort B explored same-day administration of NKTR-262 at the RP2D (3.84 mg) and bempegaldesleukin (0.006 mg/kg) q3w plus nivolumab (360 mg) q3w, starting in Cycle 1.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 NKTR-262 (0.03 mg) + Bempegaldesleukin (Administered Staggered) | Cohort 2 NKTR-262 (0.06 mg) + Bempegaldesleukin (Administered Staggered) | Cohort 3 NKTR-262 (0.06 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 4 NKTR-262 (0.12 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 5 NKTR-262 (0.24 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 6 NKTR-262 (0.48 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 7 NKTR-262 (0.96 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 8 NKTR-262 (1.92 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 9 NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort A NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort B NKTR-262 (3.84 mg) + Bempegaldesleukin + Nivolumab | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 4 | 4 | 4 | 3 | 8 | 14 | 14 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 2 | 2 | 2 | 1 | 3 | 3 | 8 | 10 | 8 | 43
  >=65 years | 2 | 0 | 2 | 1 | 2 | 3 | 1 | 0 | 0 | 4 | 6 | 21
Age, Continuous [Mean (Full Range); unit: years] | 66.0 [63 to 69] | 53.0 [39 to 64] | 51.5 [32 to 71] | 56.3 [39 to 73] | 57.0 [41 to 74] | 68.0 [58 to 79] | 55.3 [40 to 72] | 59.0 [58 to 61] | 49.0 [35 to 63] | 57.7 [30 to 81] | 60.3 [28 to 79] | 57.4 [28 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 1 | 2 | 2 | 1 | 0 | 5 | 4 | 7 | 26
  Male | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 3 | 10 | 7 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 3 | 3 | 4 | 2 | 3 | 4 | 4 | 3 | 8 | 13 | 13 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 3 | 8 | 11 | 14 | 59
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 3 | 4 | 4 | 4 | 3 | 8 | 14 | 14 | 64
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status
  ECOG Performance Status of 0 = Able to carry out all normal activities without restriction
  ECOG Performance Status of 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature
  Participants
    ECOG 0 | 2 | 1 | 2 | 1 | 2 | 2 | 3 | 3 | 6 | 7 | 5 | 34
    ECOG 1 | 1 | 2 | 2 | 2 | 2 | 2 | 1 | 0 | 2 | 7 | 9 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose-Limiting Toxicities (DLTS)
Description: DLTs were assessed in Cohort 1 through Cohort 9, which had dose levels of NKTR-262 as 0.03mg, 0.06mg, 0.06mg, 0.12mg, 0.24mg, 0.48mg, 0.96mg, 1.92mg, and 3.84mg in combination with bempegaldesleukin (bempeg).
  There was only 1 DLT that occurred in one of the Cohort 9 patients. Therefore, the maximum tolerated dose (MTD) of NKTR 262 was not reached.
Time Frame: The DLT window is 21 days following NKTR-262 single agent administration (Cycle 1) and an additional 9 days when combined with bempeg for staggered dosing administration (Cohorts 1 and 2), or 7 days for the same day administration (Cohort 3 and higher).
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2 NKTR-262 (0.06 mg) + Bempegaldesleukin (Administered Staggered): Phase 1 (dose escalation) Cohort 2 Patients received NKTR-262 intratumorally at 0.06 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) (administered staggered [Day 3] in Cycles 2-3).The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort B NKTR-262 (3.84 mg) + Bempegaldesleukin + Nivolumab: Cohort B explored same-day administration of NKTR-262 intratumorally at the RP2D (3.84 mg) and bempegaldesleukin IV (0.006 mg/kg) q3w plus nivolumab (360 mg) q3w, starting in Cycle 1.
Arm/Group | Cohort 1 NKTR-262 (0.03 mg) + Bempegaldesleukin (Administered Staggered) | Cohort 2 NKTR-262 (0.06 mg) + Bempegaldesleukin (Administered Staggered) | Cohort 3 NKTR-262 (0.06 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 4 NKTR-262 (0.12 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 5 NKTR-262 (0.24 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 6 NKTR-262 (0.48 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 7 NKTR-262 (0.96 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 8 NKTR-262 (1.92 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 9 NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort A NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort B NKTR-262 (3.84 mg) + Bempegaldesleukin + Nivolumab
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 3 | 4 | 3 | 7 | 11 | 13
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Objective Response Rate (ORR) Per RECIST 1.1 in Cohort A and Cohort B at Recommended Phase 2 Dose (RP2D)
Description: Objective Response Rate (ORR) per RECIST 1.1 in Cohort A and Cohort B at Recommended Phase 2 Dose (RP2D).
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 and as assessed by Blinded Independent Central Review (BICR).
Time Frame: From Cycle 1 Day 1 to 100 days after the last dose of study drug or the date for new anti-cancer therapy, whichever is earlier.
Population: safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort B NKTR-262 (3.84 mg) + Bempegaldesleukin + Nivolumab
Number analyzed (Participants) | 14 | 14
percentage of participants | 0 [0.0 to 23.2] | 14.3 [1.8 to 42.8]

ADVERSE EVENTS:
Time Frame: 4 years
Groups:
- Cohort 1 NKTR-262 (0.03 mg) + Bempegaldesleukin (Administered Staggered): Patients received NKTR-262 intratumorally at 0.03 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) (administered staggered [Day 3] in Cycles 2-3). The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort 2 NKTR-262 (0.06 mg) + Bempegaldesleukin (Administered Staggered): Patients received NKTR-262 intratumorally at 0.06 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) (administered staggered [Day 3] in Cycles 2-3).The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort 3 NKTR-262 (0.06 mg) + Bempegaldesleukin (Administered the Same Day): Patients received NKTR-262 intratumorally at 0.06 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) administered on the same day. The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort 4 NKTR-262 (0.12 mg) + Bempegaldesleukin (Administered the Same Day): Patients received NKTR-262 intratumorally at 0.12 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) administered on the same day. The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort 5 NKTR-262 (0.24 mg) + Bempegaldesleukin (Administered the Same Day): Patients received NKTR-262 intratumorally at 0.24 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) administered on the same day. The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort 6 NKTR-262 (0.48 mg) + Bempegaldesleukin (Administered the Same Day): Patients received NKTR-262 intratumorally at 0.48 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) administered on the same day. The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort 7 NKTR-262 (0.96 mg) + Bempegaldesleukin (Administered the Same Day): Patients received NKTR-262 intratumorally at 0.96 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) administered on the same day. The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort 8 NKTR-262 (1.92 mg) + Bempegaldesleukin (Administered the Same Day): Patients received NKTR-262 intratumorally at 1.92 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) administered on the same day. The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
- Cohort 9 NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day): Patients received NKTR-262 intratumorally at 3.84 mg (in Cycles 1 through 3) plus bempegaldesleukin IV at 0.006 mg/kg (starting in Cycle 2) every 3 weeks (q3w) administered on the same day. The number of patients to be enrolled per cohort was dependent the on the 3+3 study design and continued until RP2D was determined.
Arm/Group | Cohort 1 NKTR-262 (0.03 mg) + Bempegaldesleukin (Administered Staggered) | Cohort 2 NKTR-262 (0.06 mg) + Bempegaldesleukin (Administered Staggered) | Cohort 3 NKTR-262 (0.06 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 4 NKTR-262 (0.12 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 5 NKTR-262 (0.24 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 6 NKTR-262 (0.48 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 7 NKTR-262 (0.96 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 8 NKTR-262 (1.92 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort 9 NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort A NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day) | Cohort B NKTR-262 (3.84 mg) + Bempegaldesleukin + Nivolumab
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3 | 3/4 | 1/3 | 4/4 | 4/4 | 1/4 | 2/3 | 5/8 | 9/14 | 5/14
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 1/4 | 1/3 | 1/4 | 1/4 | 1/4 | 3/3 | 3/8 | 2/14 | 5/14
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 3/3 | 4/4 | 4/4 | 4/4 | 3/3 | 8/8 | 14/14 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 NKTR-262 (0.03 mg) + Bempegaldesleukin (Administered Staggered) (N=3) | Cohort 2 NKTR-262 (0.06 mg) + Bempegaldesleukin (Administered Staggered) (N=3) | Cohort 3 NKTR-262 (0.06 mg) + Bempegaldesleukin (Administered the Same Day) (N=4) | Cohort 4 NKTR-262 (0.12 mg) + Bempegaldesleukin (Administered the Same Day) (N=3) | Cohort 5 NKTR-262 (0.24 mg) + Bempegaldesleukin (Administered the Same Day) (N=4) | Cohort 6 NKTR-262 (0.48 mg) + Bempegaldesleukin (Administered the Same Day) (N=4) | Cohort 7 NKTR-262 (0.96 mg) + Bempegaldesleukin (Administered the Same Day) (N=4) | Cohort 8 NKTR-262 (1.92 mg) + Bempegaldesleukin (Administered the Same Day) (N=3) | Cohort 9 NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day) (N=8) | Cohort A NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day) (N=14) | Cohort B NKTR-262 (3.84 mg) + Bempegaldesleukin + Nivolumab (N=14)
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 NKTR-262 (0.03 mg) + Bempegaldesleukin (Administered Staggered) (N=3) | Cohort 2 NKTR-262 (0.06 mg) + Bempegaldesleukin (Administered Staggered) (N=3) | Cohort 3 NKTR-262 (0.06 mg) + Bempegaldesleukin (Administered the Same Day) (N=4) | Cohort 4 NKTR-262 (0.12 mg) + Bempegaldesleukin (Administered the Same Day) (N=3) | Cohort 5 NKTR-262 (0.24 mg) + Bempegaldesleukin (Administered the Same Day) (N=4) | Cohort 6 NKTR-262 (0.48 mg) + Bempegaldesleukin (Administered the Same Day) (N=4) | Cohort 7 NKTR-262 (0.96 mg) + Bempegaldesleukin (Administered the Same Day) (N=4) | Cohort 8 NKTR-262 (1.92 mg) + Bempegaldesleukin (Administered the Same Day) (N=3) | Cohort 9 NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day) (N=8) | Cohort A NKTR-262 (3.84 mg) + Bempegaldesleukin (Administered the Same Day) (N=14) | Cohort B NKTR-262 (3.84 mg) + Bempegaldesleukin + Nivolumab (N=14)
Fatigue (General disorders) | 2 | 3 | 2 | 1 | 3 | 2 | 3 | 1 | 4 | 8 | 6
Influenza like illness (General disorders) | 2 | 0 | 2 | 1 | 2 | 2 | 0 | 1 | 5 | 8 | 6
Pyrexia (General disorders) | 0 | 2 | 2 | 1 | 2 | 2 | 2 | 3 | 2 | 2 | 9
Chills (General disorders) | 0 | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 1 | 1 | 5
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 1 | 2
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Application site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Application site nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device related thrombosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 2 | 1 | 2 | 2 | 2 | 3 | 5 | 8 | 8
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 2 | 2 | 1 | 1 | 3 | 7 | 6
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 1 | 1 | 0 | 1 | 5 | 4 | 5
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 2 | 1 | 2 | 1 | 0 | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lip oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 0 | 3 | 1 | 0 | 3 | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 2 | 0 | 2 | 1 | 2 | 1 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 5 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Macule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 4 | 6 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 2 | 2 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1
Weight decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cortisol decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Occult blood positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 3 | 4
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 3 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blepharochalasis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Corneal opacity (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye discharge (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Open angle glaucoma (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Posterior capsule opacification (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal exudates (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device occlusion (Product Issues) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are restrictions to the PI's rights to discuss or publish trial results.

DOCUMENTS (2):
  • Study Protocol (2020-04-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT03435640/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT03435640/SAP_001.pdf